CLINICAL TRIAL: NCT01436045
Title: A Double-Blind, Placebo-Controlled Single Dose Study of the Safety and Efficacy of Glulisine on Cognitive Function and Memory in Individuals Diagnosed With Probable Mild to Moderate Alzheimer's Disease/Intranasal Insulin Study.
Brief Title: Safety and Effectiveness Study of Intranasal Insulin Glulisine on Cognitive and Memory in Mild-Mod AD Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-111
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer's Disease
Keywords: Memory; Insulin glulisine; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — insulin glulisine; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin glulisine (Experimental): A randomized, double-blind, placebo-controlled, cross-over designed - all subject will receive intervention (insulin glulisine) and placebo (saline) during separate visits.
  Interventions: Drug: Insulin glulisine
- Saline (Placebo Comparator): A randomized, double-blind, placebo-controlled, cross-over designed - all subject will receive intervention (insulin glulisine) and placebo (saline) during separate visits.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Insulin glulisine — Single treatment, 20 IU/Intranasal (.1ml/10 units Intranasally in each nostril)
  Other Names: Apidra
  Arms: Insulin glulisine
Drug: Saline — Single treatment,(saline) 20 IU/Intranasal (.1ml/10units intranasally in each nostril)
  Other Names: salt water
  Arms: Saline

SUMMARY:
The purpose of this study is to investigate the effect of the rapidly acting intranasal insulin derivative (glulisine) on memory and cognition in 12 patients suffering from mild-moderate Alzheimer's Disease (AD) using a double-blind placebo-controlled single dose study. This study will further assess safety of insulin glulisine as well as the effects of this drug on olfaction.

DETAILED DESCRIPTION:
A single center, phase II randomized, double-blind, placebo-controlled, cross-over study designed to assess the efficacy and safety of intranasally (IN) delivered insulin glulisine versus placebo in patients aged 65-85 with mild-moderate Alzheimer's Disease (AD). Twelve AD subjects (six female and six male) will be randomized to receive a single dose of either 20 IU/IN insulin glulisine or placebo using the MAD 300 device.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with a clinical diagnosis of probable AD in accordance with National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria and Dementia Rating Scale (McKhann 1984).
* Mini-Mental State Examination (MMSE) score of 18-26.
* Hachinski Ischemia Score < 4.
* Age is > 65 and <85 years
* Females must be > 2 years post-menopausal or surgically sterile.
* Must be able to speak, read and understand English in order to comply with testing of cognitive function, memory and physiology.
* Must have a dedicated family member /caregiver, able to attend all visits and report on subject's status.
* Subject and family member/caregiver have both provided fully informed written consent prior to participation. In the event that subject is legally unable to provide informed written consent due to deterioration in cognitive abilities, fully informed written consent must be provided by a legally authorized representative.
* On a stable dose (≥ 1 months) of a prescribed acetylcholinesterase inhibitor (e.g. donepezil, rivastigmine, galantamine) and/or memantine.
* A brain CT or MRI in the last 2 years compatible with the diagnosis of probable Alzheimer's Disease.
* A Clinical Dementia Rating (CDR) ranging from 1 to 2.

Exclusion Criteria:

* Medical history and/or clinically determined evidence of other central nervous system (CNS) disorders including brain tumor, active subdural hematoma, seizure disorder, multiple sclerosis dementia with Lewy bodies, vascular dementia, corticobasal syndrome, progressive supranuclear palsy, Parkinson's disease, multiple system atrophy, frontotemporal dementia, normal pressure hydrocephalus, Huntington's disease, or Jakob-Creutzfeldt disease presenting as dementia.
* Personal medical history and/or clinically determined disorders: current B12 deficiency, positive syphilis serology, chronic sinusitis or any untreated thyroid disease, significant head trauma, or history of difficulty with smell and/or taste prior to AD diagnosis.
* Diagnosis with any form of diabetes mellitus, actively takes insulin, or has HbA1c > 6.1 % at screening.
* Personal history of any of the following: moderate to severe pulmonary disease, congestive heart failure, significant cardiovascular and/or cerebrovascular events in previous 6 months, condition known to affect absorption, distribution, metabolism, or excretion of drugs such as any hepatic, renal or gastrointestinal disease or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by Investigator.
* Heavy smoker (defined as smoking half a pack or more per day in the last 10 years prior to entry in the study).
* Personal history of any psychiatric illness, except major depressive disorder (according to Diagnostic and Statistical Manual (DSM)-IV TR) currently in remission or stable with treatment for > 2 years, or any other psychiatric condition that inclusion would pose a safety risk to the subject as determined by Investigator. Patients with active depression (Geriatric Depression Score>9) are excluded from the study.
* Currently taking any medications, herbals and food supplements that are determined by Investigator to interfere with procedural testing of cognitive function as well as ensure study safety.
* Recent change (< 1 months) in prescribed acetylcholinesterase inhibitor (e.g. donepezil, rivastigmine, galantamine) or memantine.
* Current or recent drug or alcohol abuse or dependence defined by DSM-IV TR.
* Systolic blood pressure > 160 or < 90 mmHg or diastolic blood pressure > 100 or < 60 mmHg at Screening.
* Screening laboratory results that are medically relevant and which would pose a safety risk to the subject as determined by Investigator.
* Participation in any other research study at least 3 months prior to this study.
* Insulin allergy.
* History of significant traumatic brain injury
* History of acute and chronic rhinitis and/or sinusitis.
* Legally unable to provide informed written consent due to deterioration in cognitive abilities.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Specialty Center - Center for Dementia & Alzheimer's Care, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Glulisine, Then Placebo: A randomized, double-blind, placebo-controlled, cross-over designed - all subject will receive intervention (insulin glulisine) and placebo (saline) during separate visits.
  Insulin glulisine (5 minutes), Washout (1 week), Placebo (5 minutes)
  Insulin glulisine: Single treatment, 20 IU/Intranasal (.1ml/10 units Intranasally in each nostril)
  Placebo: Single treatment,(saline) 20 IU/Intranasal (.1ml/10units intranasally in each nostril)
- Placebo, Then Insulin Glulisine: A randomized, double-blind, placebo-controlled, cross-over designed - all subject will receive intervention (insulin glulisine) and placebo (saline) during separate visits.
  Placebo (5 minutes), Washout (1 week), Insulin Glulisine (5 minutes)
  Insulin glulisine: Single treatment, 20 IU/Intranasal (.1ml/10 units Intranasally in each nostril)
  Placebo: Single treatment,(saline) 20 IU/Intranasal (.1ml/10units intranasally in each nostril)
Period: Overall Study
Arm/Group | Insulin Glulisine, Then Placebo | Placebo, Then Insulin Glulisine
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Partipants: Participants who received either intranasal glulisine (0.10 milliliter (mL) in each nostril, 20 IU total) or placebo (0.10 mL in each nostril) at the 2nd or 3rd study visit.
Arm/Group | All Study Partipants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — MMSE scale is 0 to 30. Lower scores indicate more severe cognitive impairment. Higher scores (27-30) indicate normal cognition.
  units on a scale | 22.17 (2.62)
University of Pennsylvania Smell Inventory Test (UPSIT) [Mean (Standard Deviation); unit: units on a scale] — UPSIT is used to test the function of an individual's olfactory system. The first 20 items (out of 40) were used. Range of 0-20. Lower scores indicate a lower functioning olfactory system. Higher scores indicate normal olfactory functioning.
  units on a scale | 11.8 (2.52)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Performance
Description: The results are presented as a mean number of correct responses for each cognitive assessment.
  For each of these, a lower number correct is indicative of a higher cognitive deficit.
  Ranges are as follows: RBANS List Learning (0-40), RBANS Story Memory (0-24), RBANS Figure Copy (0-20), RBANSLine Orientation (0-20), RBANS Semantic Fluency (0-unlimited), RBANS List Recall (0-10), RBANS List Recognition (0-20), RBANS Story Recall (0-12), RBANS Figure Recall (0-20), Digit Span Forward (0-16), Digit Span Backward (0-16), Boston Naming (0-15).
Time Frame: 20 minutes post-intranasal administration
Measure: Mean (Standard Error); unit: mean total correct responses
Groups:
- Post-Insulin Glulisine: Results of cognitive assessment after intranasal treatment with Insulin Glulisine.
- Post-Placebo: Results of cognitive assessment after intranasal treatment with Placebo.
Arm/Group | Post-Insulin Glulisine | Post-Placebo
Number analyzed (Participants) | 12 | 12
mean total correct responses
  RBANS List Learning | 15.92 (1.32) | 16.67 (2.02)
  RBANS Story Memory | 8.58 (1.17) | 8.41 (1.55)
  RBANS Figure Copy | 16.58 (0.98) | 16.92 (3.42)
  RBANS Line Orientation | 14.25 (0.97) | 12.25 (1.38)
  RBANS Semantic Fluency | 12.25 (1.38) | 12.5 (1.75)
  RBANS List Recall | 0.83 (0.42) | 1.0 (0.51)
  RBANS List Recognition | 14.92 (0.69) | 14.75 (0.97)
  RBANS Story Recall | 2.12 (0.96) | 2.33 (0.90)
  RBANS Figure Recall | 4.83 (1.84) | 4.92 (1.59)
  Digit Span Forward | 9.42 (0.50) | 9.0 (0.44)
  Digit Span Backward | 5.58 (0.45) | 5.75 (0.49)
  Boston Naming Test | 11.75 (1.05) | 11.75 (1.10)
Statistical Analysis 1: Comparison: Post-Insulin Glulisine vs Post-Placebo; Response to intranasal Insulin Gluiline [(result post-insulin - result post-placebo)/(result post-placebo)] x 100%; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — RBANS Line Orientation; Percent Change = -15.7, Standard Error of Mean 7.0 — Response to intranasal Insulin Glulisine [(result post-insulin - result post-placebo)/(result post-placebo)] x 100%

2. Secondary Outcome: Olfactory Function
Description: The Sniff Magnitude Test (SMT) measures olfactory function not influenced by cognitive problems (minimal dependence on language, cognitive ability, memory, and odor naming ability). Sniff magnitude ratios are calculated as a ratio of sniff magnitudes (area under the sniff curve). Lower sniff magnitude ratios indicate more impairment.
  [average sniff magnitude of malodor/average sniff magnitude to a null odor]
Time Frame: 60 minute post intranasal administration
Measure: Mean (Standard Error); unit: ratio of area under the sniff curve
Groups:
- Post Placebo: Results of cognitive assessment after intranasal treatment with Placebo.
Arm/Group | Post-Insulin Glulisine | Post Placebo
Number analyzed (Participants) | 12 | 12
ratio of area under the sniff curve | 2.5 (0.15) | 2.33 (0.19)

3. Primary Outcome: Trails B - Seconds
Description: The results are presented as the number of seconds to complete Trails B. For each of these, a higher number of seconds is indicative of a higher cognitive deficit.
Time Frame: 20 minutes post-intranasal administration
Measure: Mean (Standard Error); unit: mean seconds
Arm/Group | Post-Insulin Glulisine | Post-Placebo
Number analyzed (Participants) | 12 | 12
mean seconds | 166.83 (20.82) | 177.25 (21.65)

4. Primary Outcome: Trails B - Errors
Description: The results are presented as the mean sum of the errors during the Trails B assessment For each of these, a higher number of errors is indicative of a higher cognitive deficit.
Time Frame: 20 minutes post-intranasal administration
Measure: Mean (Standard Error); unit: mean number of errors
Arm/Group | Post-Insulin Glulisine | Post-Placebo
Number analyzed (Participants) | 12 | 12
mean number of errors | 1.17 (0.27) | 2.08 (0.31)
Statistical Analysis 1: Comparison: Post-Insulin Glulisine vs Post-Placebo; Difference in errors [result post-insulin - result post-placebo]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.92, Standard Error of Mean 0.26

ADVERSE EVENTS:
Groups:
- All Study Partipants: Participants who received either intranasal glulisine (0.10 mL in each nostril, 20 IU total) or placebo (0.10 mL in each nostril) at the 2nd or 3rd study visit.
Arm/Group | All Study Partipants
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes